CLINICAL TRIAL: NCT03012035
Title: The Role of Treatment Expectation in Exposure Training With Spider Fearful Participants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: SPFE 2017
Record Dates: First submitted 2016-12-21; First posted 2017-01-06 (Estimated); Last update posted 2018-03-21 (Actual); Status verified 2018-03

CONDITIONS: Phobic Disorders
Keywords: psychotherapy; exposition; spider fear; expectation
MeSH Terms: conditions — Phobic Disorders; Arachnophobia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): Before participants undergo the exposure training their expectation of treatment efficacy is manipulated with different information regarding the following treatment. The experimental group will get positive treatment expectations induced with the accurate information, that exposure training refers to the gold standard in psychotherapy to reduce spider fear (= open administration of treatment).
  Interventions: Other: positive treatment expectations
- comparator group (Other): The comparator group will get neutral expectations regarding treatment outcome. To induce neutral treatment expectations about the following exposure training, it is necessary to tell them they are in the comparator group and that they will receive a comparator condition exposure training for diagnostic purposes only (= hidden administration of treatment).
  Interventions: Other: neutral treatment expectations

INTERVENTIONS:
Other: positive treatment expectations — Before participants undergo the exposure training their expectation of treatment efficacy is manipulated with different information regarding the following treatment. The experimental group will get positive treatment expectations induced with the accurate information, that exposure training refers to the gold standard in psychotherapy to reduce spider fear (= open administration of treatment).
  Arms: experimental group
Other: neutral treatment expectations — The comparator group will get neutral expectations regarding treatment outcome. To induce neutral treatment expectations about the following exposure training, it is necessary to tell them they are in the comparator group and that they will receive a comparator condition exposure training for diagnostic purposes only (= hidden administration of treatment).
  Arms: comparator group

SUMMARY:
This study evaluates the role of treatment success expectation in spider fearful individuals on the actual treatment success. Half of participants will have positive treatment success expectations, while the other half will have neutral treatment outcome expectations.

DETAILED DESCRIPTION:
The investigator plan to conduct a randomized, single blind study with two parallel groups. Both groups undergo the same standardized psychotherapeutic intervention, i.e. exposure training. All participants will receive the same exposure training in groups of maximum three participants of the same study group. The two study groups only differ regarding the induced treatment expectations towards the effects of the exposure training. While the experimental group will get an open administration of treatment and be informed in order to have a positive treatment expectation, the comparator group will receive a hidden administration of treatment and get neutral information, thus treatment expectations will be neutral. Study members conducting the exposure training with the participants will not be aware of the allocation of the study participants. Study participants will be informed about the aim of the allocated condition, but they will be blind to the aim of the study in order to induce the specific expectation. Differences in treatment outcomes are compared between both groups to investigate the association with treatment expectation.

ELIGIBILITY:
Inclusion Criteria:

* good knowledge of German language
* fulfilling criteria A-E and G for specific phobia according to Diagnostic and Statistical Manual of Mental Disorders (DSM)-V (fulfilling criteria F is not an inclusion criteria)

  * marked fear or anxiety about spiders
  * spiders almost always provoke immediate fear or anxiety
  * spiders are actively avoided or endured with intense fear or anxiety
  * the fear or anxiety is out of proportion to the actual danger posed by spiders
  * the fear, anxiety, or avoidance is persistent, typically lasting for 6 months or more
  * the disturbance is not better explained by the symptoms of mental disorders as agoraphobia, obsessive-compulsive disorder, posttraumatic stress disorder, separation anxiety or social anxiety disorder

Exclusion Criteria:

* acute or chronic psychiatric disorder
* currently in psychological or psychiatric treatment
* knowledge of exposure training

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2017-05-18 (Actual); Primary Completion 2018-03-12 (Actual); Study Completion 2018-03-12 (Actual)

PRIMARY OUTCOMES:
Change in subjective anxiety assessed by questionnaire | Baseline, Pre exposition, Post exposition, Recovery; time between baseline and recovery approximately lasts 21 days
  assessment of change in subjective anxiety by questionnaire at selcted time points

CONTACTS AND LOCATIONS:
Overall Officials: Jens Gaab, Prof. Dr., Principal Investigator — Department of Clinical Psychology and Psychotherapy University of Basel
Locations (1):
- Department of Clinical Psychology and Psychotherapy University of Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No